CLINICAL TRIAL: NCT00281385
Title: Health and Psychological Outcomes of Lifestyle Versus Traditional Physical Activity- Study 1
Brief Title: Health and Psychological Outcomes of Lifestyle Versus Traditional Physical Activity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-0422-02; CIHR
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Sedentary Behaviour; Adherence; Traditional Exercise; Lifestyle Exercise
Keywords: adherence; lifestyle; exercise; pedometer; training
MeSH Terms: conditions — Motor Activity

INTERVENTIONS:
Behavioral: traditional vs. lifestyle exercise

SUMMARY:
This study is a comparison of the traditional prescription versus the lifestyle exercise prescription in sedentary adults over 6 months. Biological and psychological parameters will be assessed over the 6 month study. Biological indicators will be assessed pre and post including body composition, muscular strength, endurance, and flexibility, aerobic fitness, and blood tests. Psychological parameters will be assessed pre, mid, and post including self-efficacy, motivation, need satisfaction, physical self-description, leisure-time exercise, as well as all constructs from the thepry of planned behaviour.

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years old
* exercise less than twice per month in the preceeding 6 months
* physician consent to participate

Exclusion Criteria:

* health problems
* exercise more than twice per month in the preceeding 6 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Rodgers, PhD., Principal Investigator — University of Alberta; Gordon J Bell, PhD, Principal Investigator — University of Alberta; Kerry Courneya, PhD, Principal Investigator — University of Alberta; Vicki J Harber, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada